CLINICAL TRIAL: NCT06621355
Title: HemoNIRS: Un Cambio De Paradigma En El Proceso De Rehabilitación Musculoesquelética De Lesiones De Ligamento Cruzado Anterior Mediante Dispositivos NIRS En Deportistas Que Realizan Deportes Cíclicos
Brief Title: HemoNIRS: a Paradigm Shift in the Process of Musculoskeletal Rehabilitation of ACL Injuries in Cyclic Sports Athletes.
Status: Not yet recruiting | Type: Observational
Sponsor: Universitat de Lleida (Other)
Responsible Party: Principal Investigator, Xisco Verdejo, PhD Student and Associate Professor, Universitat de Lleida
Other Study IDs: HemoNIRS-LCA
Record Dates: First submitted 2024-09-25; First posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: ACL - Anterior Cruciate Ligament Rupture; ACL Injury; Hemodynamics; Oxygen Consumption Based Assessment of Hemodynamics; Exercise
Keywords: Spectroscopy, Near-Infrared; Hemodynamics; Exercise; Vascular resistance; Oxygen consumption
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries; Motor Activity | interventions — Exercise Test

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- LCA1: Patients with ACL involvement (with less than 6 months of evolution since the surgical intervention (IQ)) and are in a phase in which they can perform the incremental intervallic test either on a cycloergometer or treadmill.
  Interventions: Other: Physical fitness test: Progressive intervalic test
- LCA2: Patients who have recovered from an ACL injury for more than 2 years. And can perform the incremental intervallic test either on a cycloergometer or treadmill.
  Interventions: Other: Physical fitness test: Progressive intervalic test
- CON: Patients who have never suffered an ACL injury or involvement to date. And can also perform the test.
  Interventions: Other: Physical fitness test: Progressive intervalic test

INTERVENTIONS:
Other: Physical fitness test: Progressive intervalic test — An incremental interval test of 4' of work for 1' of rest will be performed at an individual intensity below the aerobic threshold. At the end of the rest minute, the load shall be increased slightly. In order to be as adjusted and individualised as possible, the subjective physical condition level stated by the patient during the sociodemographic data collection shall be taken as a reference for the establishment of the initial load, being a value of power (W) in cycle ergometer and speed (km/h) in treadmill. Never less than 50W or 6 km/h, respectively.
  The minimum incremental values will be 25W or 0.5km/h until you are unable to complete a full interval. An incomplete interval shall also be recorded and analysed.
  During the one minute rest period, as will have been well emphasised during the explanation of the test, no part of the body may be moved at all, so at the end of the 4 minutes of work, the evaluator will count down for the patient to get ready and remain stil
  Other Names: Physical fitness test

SUMMARY:
Muscle haemodynamics has so far been assessed using at most 2-3 near-infrared spectroscopy devices on isolated muscles and without correlating variables. At the same time, research on musculoskeletal pathologies is limited, and there are no studies that analyse the haemodynamic changes that occur when the anterior cruciate ligament (ACL) is injured and whether these changes last over time. The aim of the study is to monitor and evaluate the physiological changes produced by ACL injury on muscle performance using non-invasive near-infrared spectroscopy (NIRS) devices in trained athletes. This descriptive cross-sectional observational multicentre multicentre study, with Balearic Islands ethics committee IB 5585/24PI, will include males aged 18-65 years who have undergone ACL surgery, divided into 3 groups that: have an evolution of less than 6 months (ACL1), more than 2 years since the surgical intervention and are already practising normal physical-sports activities (ACL2) and the control group (CON) that has never suffered an ACL affectation to date. The 3 groups will perform an incremental intervallic test (4:1) on a cycloergometer or treadmill (according to the specificity of their sport), where different muscular haemodynamic variables will be assessed using 12-24 NIRS devices. The main study variables will be the muscular haemodynamic values of each muscle analysed and their correlation between them: muscular oxygen saturation, absolute capillary haemoglobin, loaded and unloaded with oxygen and relative muscular haemoglobin blood flow, loaded and unloaded with oxygen. Secondary variables will be heart rate, socio-demographic variables (age, toxic habits, injury and sports history) and subjective perception of effort (RPE-20).

DETAILED DESCRIPTION:
This study aims to investigate the physiological changes occurring in the musculoskeletal system during the rehabilitation process of ACL injuries using Near-Infrared Spectroscopy (NIRS) technology. This study explores how NIRS devices can monitor muscle hemodynamics during specific rehabilitation exercises, providing real-time insights into the muscle performance and recovery status of patients. The research focuses on athletes who have undergone ACL surgery, categorizing them into different groups based on the time since their surgical intervention (<6 months post-surgery and >2 years post-surgery) compared to a control group that has no history of ACL injury. The study follows a multicenter, observational, cross-sectional, descriptive design and is conducted across multiple healthcare centers, including Físic Espai de Salut Integral, Centre Re3MOVE, MET Salut, Hospital Universitari Son Espases, and San Juan de Déu Palma-Inca. These centers have been selected to ensure a diverse and representative sample of participants, focusing on sports rehabilitation specialists and integrating technology for evaluating functional recovery and muscle performance during rehabilitation.

The participants include male athletes aged 18 to 65 years, who are divided into three distinct groups. Group 1 (LCA1) consists of athletes who have undergone ACL surgery within the last 6 months and are currently undergoing rehabilitation. Group 2 (LCA2) consists of athletes who have had ACL surgery more than 2 years ago and have returned to their normal sporting activities. Group 3 (control group) consists of healthy athletes with no history of ACL injury. The primary objective of the study is to evaluate the physiological and hemodynamic changes in muscle function during rehabilitation and to establish how these changes persist over time. Additionally, the study aims to identify residual physiological limitations in the musculoskeletal system post-rehabilitation and surgery. The specific muscles of interest include the rectus femoris, vastus lateralis, gluteus maximus, hamstrings, and other stabilizing muscles in both the lower and upper body, depending on the mode of exercise used in the evaluation.

NIRS technology, which is non-invasive, will be employed to monitor muscle oxygen saturation (SmO2), total hemoglobin concentration (ThB), oxygenated hemoglobin (O2Hb), and deoxygenated hemoglobin (HHb) in real time. These measures will allow the researchers to assess the muscle's oxidative capacity, blood flow, and overall performance during rehabilitative exercises. The tests will be conducted using a cycle ergometer or treadmill, depending on the participant's sport, and will follow an intervallic incremental protocol (4 minutes of work followed by 1 minute of rest), increasing the workload incrementally until the participant reaches their maximum capability.

The methodology incorporates the use of 12 to 24 portable NIRS devices attached to the participants' muscles, allowing for simultaneous, real-time monitoring of muscle hemodynamics during exercise. The devices will be linked to a central software system (PeriPedal), which will collect and analyze the data, providing feedback to the researchers about muscle performance. Secondary outcomes of the study include heart rate monitoring, body composition (using bioimpedance and skinfold thickness measurements), and subjective perception of exertion using the RPE-20 scale. Sociodemographic data, such as age, injury history, and physical activity levels, will also be collected to contextualize the findings.

This study will adopt a pragmatic approach by incorporating the NIRS technology into routine clinical practice, aiming to create a more holistic understanding of muscle hemodynamics during ACL rehabilitation. The primary hypothesis of the study is that ACL injuries produce measurable changes in muscle hemodynamics that persist over time, even after successful rehabilitation. By identifying the factors that limit muscle performance in real-time, the study seeks to provide clinicians with new tools to tailor rehabilitation programs more effectively and reduce the incidence of recurrent injuries.

The findings from this study have the potential to transform the way musculoskeletal injuries are managed, particularly in terms of rehabilitation strategies and monitoring techniques. The study also aims to contribute to the broader understanding of how muscle performance is influenced by ACL injuries and rehabilitation, ultimately improving patient outcomes in both clinical and athletic settings.

In conclusion, the HemoNIRS project is an innovative approach to understanding the physiological and hemodynamic changes in the musculoskeletal system following ACL injuries, providing real-time data that can be used to optimize rehabilitation processes and enhance overall muscle performance.

ELIGIBILITY:
General inclusion criteria

* Men aged 18 to 65
* An adipose layer of <2 cm in areas of NIRS placement, assessed with a plicometer
* Understand written, read and spoken Spanish, English or Catalan.

General exclusion criteria

* Having any cardio-metabolic, hormonal, neurological or other comorbidities that could affect participation in the study (e.g. severe mental illness, end-stage disease).

Eligibility criteria (LCA1 group)

* Regular athlete with training and/or competition >3 days/wk prior to injury.
* ACL injury <6 months after surgery.
* Able to perform an incremental intervallic test on a cycloergometer or treadmill.

Eligibility criteria (LCA2 group)

* Regular athlete with training and/or competition >3 days a week.
* ACL injury >2 years after surgery.
* Able to perform an incremental intervallic test on a cycloergometer or treadmill.

Eligibility criteria (CON group)

* Regular athlete with training and/or competition >3 days a week.
* Never suffered an ACL injury in any knee - Able to perform incremental intervallic test on cycleergometer or treadmill.

All the groups exclusion criteria

- Incapacitating pain that prevents assessment

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The sample, which will be selected by convenience, will be made up of participants who have a diagnosis of ACL involvement and who have undergone surgery (total or partial), either recently or have had an injury in previous years, may be recruited to participate in the study. Healthy, physically active patients who have never had an ACL injury will also be recruited.
  The sample will initially come from the Físic Espai de Salut Integral, Centre Re3MOVE, MET Salut, Hospital Universitari Son Espases (HUSE) and San Juan de Déu Palma-Inca centres. Other private and public physiotherapy, rehabilitation and recovery centres, as well as private entities (clubs, federations, associations and organisations) that may contain participants susceptible to being included in the study, are expected to be included as they are accepted by the respective research commissions.
Sampling Method: Non-Probability Sample
Enrollment: 129 (Estimated)
Dates: Start 2024-12-02 (Estimated); Primary Completion 2025-11-30 (Estimated); Study Completion 2026-12-02 (Estimated)

PRIMARY OUTCOMES:
Muscular Oxygen Saturation (SmO2 - %) | From the start of the test up to 3 minutes after the end of the test
  Percentage of haemoglobin + myoglobin at muscle capillary level loaded with oxygen
Absolute Capillary Haemoglobin (ThB - g/dL) | From the start of the test up to 3 minutes after the end of the test
  grams of haemoglobin + myoglobin loaded and unloaded with oxygen divided by decilitres of blood taken up by the devices in the muscle capillaries
Oxygen-loaded capillary haemoglobin (O2HHb - g/dL) | From the start of the test up to 3 minutes after the end of the test
  grams of haemoglobin + oxygen-loaded myoglobin divided by the decilitres of blood taken up by the devices in the muscle capillaries
Capillary Haemoglobin Oxygen Depleted (HHb - g/dL) | From the start of the test up to 3 minutes after the end of the test
  grams of haemoglobin + oxygen-loaded myoglobin divided by the decilitres of blood taken up by the devices in the muscle capillaries
Blood Flow of Relative Muscle Haemoglobin (ThBBF - g/dL/min) | From the start of the test up to 3 minutes after the end of the test
  relative value of haemoglobin blood flow per unit time circulating in the muscle capillary when heart rate values are added.
Blood Flow of Oxygen Loaded Relative Muscle Haemoglobin (O2HHbBF - g/dL/min) | From the start of the test up to 3 minutes after the end of the test
  Relative value of oxygen-loaded haemoglobin blood flow per unit time circulating in the muscle capillary when heart rate values are added.
Blood Flow of Oxygen Discharged Relative Muscle Haemoglobin (HHbBF - g/dL/min) | From the start of the test up to 3 minutes after the end of the test
  Relative value of the blood flow of oxygen discharged haemoglobin per unit time circulating in the muscle capillary when heart rate values are added.

SECONDARY OUTCOMES:
Heart Rate (ppm) | From the start of the test up to 3 minutes after the end of the test
  will be monitored at all times through the use of a heart rate monitoring strap (Garmin HRM-ProTm Plus) which will transmit the constants via Bluetooth to the head unit.
Subjective perception of effort (RPE-20) | From the start of the test up to 3 minutes after the end of the test. At the end of each quarter minute of test work, during the one minute rest period, the patient will be asked his or her RPE.
  Central and local (leg) fatigue shall be assessed just before the start of the test, at the rest period of each interval, at the end of the test and at 1 and 3 minutes after the end of the test. Data shall be recorded directly into the storage software using the Borg scale.
Anthropometry and adiposity indicators: height | The following variables will only be recorded once, at the beginning of the study, mainly to check that the eligibility criteria are met and to determine at a descriptive statistical level the normality and homogeneity of the sample.
  height (m)
Anthropometry and adiposity indicators: weight | The following variables will only be recorded once, at the beginning of the study, mainly to check that the eligibility criteria are met and to determine at a descriptive statistical level the normality and homogeneity of the sample.
  weight (kg).
  In addition to height, BMI (kg/m2) will also be taken.body mass index (BMI) (kg/m2)
Anthropometry and adiposity indicators: skinfolds | The following variables will only be recorded once, at the beginning of the study, mainly to check that the eligibility criteria are met and to determine at a descriptive statistical level the normality and homogeneity of the sample.
  The amount of subcutaneous adipose tissue shall be measured by skinfold assessment. The skinfolds (mm) by using a plicometer in the bicipital, tricipital, suprailiac, thigh, leg and in those areas where a NIRS device will be placed to ensure that there is a fat layer <2cm
Socio-demographic variables | To be registered only once, before the valuation.
  Age and date of birth (month/year), toxic habits, injury history (when was the last injury and of what type, and the history of most significant injuries and/or incidences), sports history (what individual or group sport they do, the dominant arm and/or leg, the sports history of their career with the time spent), physical practice in the last 48-72 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Francesc Valenzuela-Pascual, PhD, Study Director — Universitat de Lleida; Oriol Martínez-Navarro, PhD, Study Director — Universitat de Lleida

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: SAP, ICF